CLINICAL TRIAL: NCT03566316
Title: Randomized, Double-blind, Multi-center Phase III Clinical Trial to Evaluate the Efficacy and Safety of Telmisartan/Amlodipine and Rosuvastatin Co-administration in Hypertensive Patients With Hyperlipidemia
Brief Title: Efficacy/Safety of Telmisartan/Amlodipine/Rosuvastatin in Hypertensive Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ID-TAR-301
Record Dates: First submitted 2018-06-11; First posted 2018-06-25 (Actual); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Hypertension With Hyperlipidemia
MeSH Terms: interventions — telmisartan amlodipine combination; Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telmisartan/Amlodipine+Rosuvastatin (Experimental): Telmisartan/Amlodipine 40/5mg 2tab., Rosuvastatin 20mg1tab. and Telmisartan placebo 1tab.
  Interventions: Drug: Telmisartan/Amlodipine; Drug: Rosuvastatin
- Telmisartan/Amlodipine (Active Comparator): Telmisartan/Amlodipine 40/5mg 2tab., Rosuvastatin placebo 1tab. and Telmisartan placebo 1tab.
  Interventions: Drug: Telmisartan/Amlodipine
- Telmisartan +Rosuvastatin (Active Comparator): Telmisartan/Amlodipine placebo 2tab., Rosuvastatin 80mg 1tab. and Telmisartan 20mg 1tab.
  Interventions: Drug: Rosuvastatin; Drug: Telmisartan

INTERVENTIONS:
Drug: Telmisartan/Amlodipine
  Arms: Telmisartan/Amlodipine; Telmisartan/Amlodipine+Rosuvastatin
Drug: Rosuvastatin
  Arms: Telmisartan +Rosuvastatin; Telmisartan/Amlodipine+Rosuvastatin
Drug: Telmisartan
  Arms: Telmisartan +Rosuvastatin

SUMMARY:
A Randomized, Double-blind, Multi-center Phase III Clinical Trial to Evaluate the Efficacy and Safety of Telmisartan/Amlodipine and Rosuvastatin Co-administration in Hypertensive Patients with Hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

1. 19 years old or above
2. Patients who confirmed essential hypertension with Hyperlipidemia or use of drugs at Visit 1 (sit systolic blood pressure ≥ 140mmHg, LDL-Cholesterol ≥ 100mg/dL)
3. Patients who can stop the treatment of anti-hypertensive/anti-hyperlipidemic drugs in the opinion of the investigator
4. Test results showing the following values at screening time (Visit 2) : sit systolic blood pressure >140mmHg
5. Test results showing the following values at screening time (Visit 2) : 100< LDL-Cholesterol <250
6. Patients who agreed to participate in the trial

Exclusion Criteria:

1. Severe hypertension patients(systolic blood pressure ≥ 180 mm Hg or diastolic blood pressure ≥ 110 mm Hg)

   -The change of mean sit systolic blood pressure ≥ 20 mmHg or sit diastolic blood pressure ≥ 10 mmHg on target arm between 1st and 2nd measurement
2. LDL-Cholesterol > 250 mg/dL or triacylglycerol ≥ 400 mg/dL at screening time(Visit 1)
3. Patients with postural hypotension who have sign and symptom
4. Patients with secondary blood pressure(for example,aortic coarctation, hyperaldosteronism, renal artery stenosis, Cushing's syndrome, pheochromocytoma, Polycystic Kidney Diseases)
5. Patients with congestive heart failure(New York Heart Association class III~IV)
6. Patients with history of acute coronary syndrome or underwent revascularization (percutaneous transluminal coronary angioplasty or Coronary Artery Bypass Graft surgery ) within 6 months
7. Patients who have severe ventricular tachycardia, atrial fibrillation, atrial flutter or clinically significant arrhythmia
8. Causes of hemodynamic disorder or structural heart defect such as valvular heart disease
9. Patients who have history of cerebrovascular disease as cerebral infarction, cerebral hemorrhage within 6 months prior to study entry
10. Patients with primary aldosteronism
11. Patients with severe ocular disorders
12. Patients with autoimmune disease
13. Patients with any chronic inflammation disease needed to chronic inflammation therapy
14. Patients with uncontrolled diabetes Mellitus with HbA1c > 9% or thyroid diseases(TSH ≥ 1.5 X ULN)
15. Patients who have a history of myopathy or rhabdomyolysis
16. Patients who have 3 times of upper limit of normal range of muscle enzyme (creatinine kinase, CK)
17. History of malignant tumor including leukemia, lymphoma within 5 years
18. Patients with one kidney
19. Patients with biliary obstructive disorder
20. Patients with clinically significant electrolyte disturbance
21. Continued serum potassium concentration abnormal status (<3.5mEq/L or >5.5mEq/L)
22. Patients with sodium ion or body fluid is depleted and not able to correct
23. Patients with clinically significant liver/renal disease
24. Patients with digestive diseases that may affect the absorption or history in gastrointestinal surgery
25. Patients who are dependent on drugs or alcohol
26. Pregnancy, breast-feeding, or child-bearing potential Patients
27. Patients with hypersensitivity to telmisartan or other angiotensin II receptor blockers
28. Patients with hypersensitivity to Amlodipine or other dihydropyridine drugs
29. Patients with history of Myotoxicity to other 3-hydroxy-methyl glutaryl-coenzyme A reductase inhibitor or fibrate
30. Patients who are unable to stop taking prohibited drugs to combination during study period
31. Patients who have galactose intolerance
32. Patients taking other clinical trial drugs within 30 days from the time of visit for screening
33. Patients that is not eligible to participate at the discretion of study investigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2015-11-24 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2017-06-16 (Actual)

PRIMARY OUTCOMES:
Percentage of change in LDL-Cholesterol | From baseline at week 8
  Telmisartan/Amlodipine/Rosuvastatin versus Telmisartan/Amlodipine
The change of sitting systolic blood pressure | From baseline at week 8
  Telmisartan/Amlodipine/Rosuvastatin versus Telmisartan/Rosuvastatin

SECONDARY OUTCOMES:
Percentage of change in LDL-Cholesterol | From baseline at week 4
Percentage of change in HDL-Cholesterol, total Cholesterol, Triglyceride, Apolipoprotein B | From baseline at week 4 and 8
The change of HDL-Cholesterol/LDL-Cholesterol ratio | From baseline at week 4 and 8
The change of total cholesterol/HDL-Cholesterol ratio | From baseline at week 4 and 8
Percentage of patients reaching treatment goals according to National Cholesterol Education Program-Adults Treatment Panel III Guideline | From baseline at week 4 and 8
The change of sitting diastolic blood pressure | From baseline at week 4 and 8
Percentage of patients reaching treatment goals according to Joint National Committee VIII Guideline | From baseline at week 4 and 8

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim TS, Rha SW, Kim SY, Park DG, Sung KC, Yoon MH, Kim KH, Lee HC, Kim WS, Kim YJ, Ahn JC, Rhee MY, Cha DH, Yoo BS, Park SH, Yoo KD, Jeon DW, Yoon YW, Cho SK, Oh YS. Efficacy and Tolerability of Telmisartan/Amlodipine and Rosuvastatin Coadministration in Hypertensive Patients with Hyperlipidemia: A Phase III, Multicenter, Randomized, Double-blind Study. Clin Ther. 2019 Apr;41(4):728-741. doi: 10.1016/j.clinthera.2019.02.013. Epub 2019 Mar 21. PMID 30904178